CLINICAL TRIAL: NCT05372588
Title: A Multi-Part, Phase 3, Randomized, Observer Blinded Study to Evaluate the Safety and Immunogenicity of Omicron Subvariant and Bivalent SARS-CoV-2 rS Vaccines in Adults Previously Vaccinated With Other COVID-19 Vaccines
Brief Title: Phase 3 Boosting Study for the SARS-CoV-2 rS Variant Vaccines
Acronym: COVID-19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novavax (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2019nCoV- 311
Record Dates: First submitted 2022-05-09; First posted 2022-05-12 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: COVID-19; SARS CoV 2 Infection
Keywords: Coronavirus
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — NVX-CoV2373 adjuvated lipid nanoparticle

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (8):
- Group A (NVX-CoV2515 ) (Experimental): 1 intramuscular (IM) injection of NVX-CoV2515 of 0.5 mL injection volume on Day 0.
  Interventions: Drug: NVX-CoV2515
- Group B (NVX-CoV2373 ) (Experimental): 1 intramuscular (IM) injection of NVX-CoV2373 of 0.5 mL injection volume on Day 0.
  Interventions: Drug: NVX-Cov2373
- Group C (NVX-CoV2515 ) (Experimental): 1 intramuscular (IM) injection of NVX-CoV2515 of 0.5 mL injection volume on Day 0.
  Interventions: Drug: NVX-CoV2515
- Group D (NVX-CoV2373) (Experimental): 1 intramuscular (IM) injection of NVX-CoV2373 of 0.5 mL injection volume on Day 0.
  Interventions: Drug: NVX-Cov2373
- Group E (BA.1 Bivalent Vaccine) (Experimental): 1 intramuscular (IM) injection of Bivalent Vaccine (NVX-CoV2373 + NVX-CoV2515) of 0.5 mL injection volume on Day 0.
  Interventions: Drug: NVX-CoV2373 + NVX-CoV2515
- Group F (NVX-CoV2540) (Experimental): 2 intramuscular (IM) injections of NVX-CoV2373 of 0.5 mL injection volume on Day 0 and on Day 90.
  Interventions: Drug: NVX-CoV2540
- Group G (NVX-CoV2373) (Experimental): 2 intramuscular (IM) injections of NVX-CoV2373 of 0.5 mL injection volume on Day 0 and on Day 90.
  Interventions: Drug: NVX-Cov2373
- Group H (NVX-CoV2373 + NVX-CoV2540) (Experimental): 2 intramuscular (IM) injections of NVX-CoV2373 of 0.5 mL injection volume on Day 0 and on Day 90.
  Interventions: Drug: NVX-CoV2373 + NVX-CoV2540

INTERVENTIONS:
Drug: NVX-CoV2515 — Intramuscular (deltoid) injection of co-formulated Omicron BA.1 SARS-CoV-2 rS vaccine with Matrix-M adjuvant (0.5 mL).
  Other Names: Omicron BA.1 SARS-CoV-2 rS /Matrix-M Adjuvant
  Arms: Group A (NVX-CoV2515 ); Group C (NVX-CoV2515 )
Drug: NVX-Cov2373 — Intramuscular (deltoid) injection of co-formulated prototype SARS-CoV-2 rS vaccine with Matrix-M adjuvant(0.5 mL).
  Other Names: SARS-CoV-2 rS/Matrix-M Adjuvant
  Arms: Group B (NVX-CoV2373 ); Group D (NVX-CoV2373); Group G (NVX-CoV2373)
Drug: NVX-CoV2373 + NVX-CoV2515 — Intramuscular (deltoid) injection of 5 µg total (2.5 µg NVX-CoV2373 + 2.5 µg NVX-CoV2515) with 50 µg Matrix-M adjuvant.
  Other Names: Prototype/BA.1 Bivalent Vaccine
  Arms: Group E (BA.1 Bivalent Vaccine)
Drug: NVX-CoV2540 — Intramuscular (deltoid) injection of co-formulated prototype SARS-CoV-2 rS vaccine with Matrix-M adjuvant(0.5 mL).
  Other Names: Omicron BA.5 SARS-CoV-2 rS /Matrix-M Adjuvant
  Arms: Group F (NVX-CoV2540)
Drug: NVX-CoV2373 + NVX-CoV2540 — Intramuscular (deltoid) injection of 5 µg total (2.5 µg NVX-CoV2373 + 2.5 µg NVX-CoV2515) with 50 µg Matrix-M adjuvant.
  Other Names: Prototype/BA.5 Bivalent Vaccine
  Arms: Group H (NVX-CoV2373 + NVX-CoV2540)

SUMMARY:
This is a Multi-Part, Phase 3, randomized, observer-blinded study to evaluate the safety and immunogenicity of booster doses of Omicron subvariant severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) recombinant (r) spike (S) protein nanoparticle vaccines (SARS-CoV-2 rS) adjuvanted with Matrix-M™ adjuvant (NVX-CoV2515 [BA.1] and NVX-CoV2540 [BA.5]) and bivalent (NVX-CoV2373 [prototype] + Omicron subvariant) SARS-CoV-2 rS vaccines (NVX-CoV2373 + NVX CoV2515 and NVX CoV2373 + NVX CoV2540) in previously vaccinated adults 18 years of age and older.

ELIGIBILITY:
Part 1

Inclusion Criteria:

To be included in this study, each individual must satisfy all the following criteria:

1. Adults ≥ 18 and ≤ 64 years of age at screening.
2. Willing and able to give informed consent prior to study enrollment and to comply with study procedures.
3. Female participants of childbearing potential (defined as any participant who has experienced menarche and who is NOT surgically sterile [ie, hysterectomy, bilateral tubal ligation, or bilateral oophorectomy] or postmenopausal [defined as amenorrhea ≥ 12 consecutive months]) must agree to be heterosexually inactive from at least 28 days prior to enrollment and through the end of the study OR agree to consistently use a medically acceptable method of contraception listed below from ≥ 28 days prior to and through the end of the study.
4. Is medically stable, as determined by the investigator (based on a review of health status, vital signs [to include body temperature], medical history, and targeted physical examination [to include body weight]). Vital signs must be within medically acceptable ranges prior to the vaccination.
5. Agrees to not participate in any other SARS-CoV-2 prevention or treatment trials for the duration of the study.
6. Have previously received 2 doses of the Moderna and/or Pfizer-BioNTech COVID-19 prototype vaccines with the last dose having been given ≥ 180 days prior to study vaccination or 3 doses of the Moderna and/or Pfizer-BioNTech COVID-19 prototype vaccines with the last dose having been given ≥ 90 days previously prior to the study vaccination.

Exclusion Criteria:

If an individual meets any of the following criteria, he or she is ineligible for this study:

1. Received COVID-19 vaccines other than Moderna and/or Pfizer-BioNTech in the past, inclusive of clinical trial COVID- 19 vaccines.
2. Participation in research involving receipt of investigational products (drug/biologic/device) within 90 days prior to study vaccination.
3. Received any vaccine ≤ 90 days prior to study vaccination, except for influenza vaccination which may be received > 14 days prior to study vaccination, or rabies vaccine which may be given if medically indicated.
4. Any known allergies to products contained in the investigational product.
5. Any history of anaphylaxis to any prior vaccine.
6. Autoimmune or immunodeficiency disease/condition (iatrogenic or congenital) requiring ongoing immunomodulatory therapy.
7. Chronic administration (defined as > 14 continuous days) of immunosuppressant, systemic glucocorticoids, or other immune-modifying drugs within 90 days prior to study vaccination.
8. Received immunoglobulin, blood-derived products, or immunosuppressant drugs within 90 days prior to the first study vaccination, except for rabies immunoglobulin which may be given if medically indicated.
9. Active cancer (malignancy) on therapy within 3 years prior to study vaccination (with the exception of adequately treated non-melanomatous skin carcinoma or lentigo maligna and uterine cervical carcinoma in situ without evidence of disease, at the discretion of the investigator).
10. Participants who are breastfeeding, pregnant, or who plan to become pregnant prior to the end of the study.
11. Suspected or known history of alcohol abuse or drug addiction within 2 years prior to the study vaccine dose that, in the opinion of the investigator, might interfere with protocol compliance.
12. Any other condition that, in the opinion of the investigator, would pose a health risk to the participant if enrolled or could interfere with evaluation of the study vaccine or interpretation of study results (including neurologic or psychiatric conditions likely to impair the quality of safety reporting).
13. Study team member or immediate family member of any study team member (inclusive of Sponsor, clinical research organization (CRO), and study site personnel involved in the conduct or planning of the study).

Part 2

Inclusion Criteria:

To be included in this study, each individual must satisfy all of the following criteria:

1. Adults and adolescents ≥ 18 years of age at screening.
2. Willing and able to give informed consent prior to study enrollment and to comply with study procedures.
3. Female participants of childbearing potential (defined as any participant who has experienced menarche and who is NOT surgically sterile [ie, hysterectomy, bilateral tubal ligation, or bilateral oophorectomy] or postmenopausal [defined as amenorrhea ≥ 12 consecutive months]) must agree to be heterosexually inactive from at least 28 days prior to enrollment and through the end of the study OR agree to consistently use a medically acceptable method of contraception listed below from ≥ 28 days prior to enrollment and through the end of the study.
4. Is medically stable, as determined by the investigator (based on review of health status, vital signs [to include body temperature], medical history, and targeted physical examination [to include body weight]). Vital signs must be within medically acceptable ranges prior to the first vaccination.
5. Agrees to not participate in any other SARS-CoV-2 prevention or treatment trials for the duration of the study.
6. Have previously received ≥ 3 doses of the Moderna and/or Pfizer-BioNTech monovalent and/or bivalent COVID-19 vaccines with the last dose having been given ≥ 90 days previously prior to first study booster.

Exclusion Criteria:

If an individual meets any of the following criteria, he or she is ineligible for this study:

1. Received COVID-19 vaccines other than Moderna and/or Pfizer-BioNTech in the past, inclusive of clinical trial COVID-19 vaccines.
2. Participation in research involving receipt of investigational products (drug/biologic/device) within 90 days prior to first study vaccination.
3. Received any vaccine ≤ 90 days prior to study vaccination, except for influenza vaccination which may be received > 14 days prior to first study vaccination, or rabies vaccine which may be given if medically indicated.
4. Any known allergies to products contained in the investigational product.
5. Any history of anaphylaxis to any prior vaccine.
6. Autoimmune or immunodeficiency disease/condition (iatrogenic or congenital) requiring ongoing immunomodulatory therapy.
7. Chronic administration (defined as > 14 continuous days) of immunosuppressant, systemic glucocorticoids, or other immune-modifying drugs within 90 days prior to first study vaccination.
8. Received immunoglobulin, blood-derived products, or immunosuppressant drugs within 90 days prior to first study vaccination, except for rabies immunoglobulin which may be given if medically indicated.
9. Active cancer (malignancy) on therapy within 3 years prior to first study vaccination (with the exception of adequately treated non-melanomatous skin carcinoma or lentigo maligna and uterine cervical carcinoma in situ without evidence of disease, at the discretion of the investigator).
10. Participants who are breastfeeding, pregnant, or who plan to become pregnant prior to the end of study.
11. Suspected or known history of alcohol abuse or drug addiction within 2 years prior to the first study vaccine dose that, in the opinion of the investigator, might interfere with protocol compliance.
12. Any other condition that, in the opinion of the investigator, would pose a health risk to the participant if enrolled or could interfere with evaluation of the study vaccine or interpretation of study results (including neurologic or psychiatric conditions likely to impair the quality of safety reporting).
13. Study team member or immediate family member of any study team member (inclusive of Sponsor, clinical research organization [CRO], and study site personnel involved in the conduct or planning of the study).
14. Participants with a history of myocarditis or pericarditis

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1340 (Actual)
Dates: Start 2022-05-25 (Actual); Primary Completion 2022-07-17 (Actual); Study Completion 2024-04-07 (Actual)

PRIMARY OUTCOMES:
Part 1: MN50 geometric mean titers (GMTs) to the Omicron BA.1 subvariant expressed as GMTs | Day 14
  Microneutralization [MN] geometric mean titers (GMTs) with an inhibitory concentration of 50% (MN50) to the Omicron BA.1 subvariant, assessed at Day 14 following initial study vaccination and analyzed by previous vaccine combination received.
Part 1: MN50 titer concentrations to the Omicron BA.1 subvariant vaccine expressed as seroresponse rates (SRRs) | Day 14
  Seroresponse rates (SRRs) (proportion of participants who achieve ≥ 4-fold increase from baseline [Day 0]) in MN50 titer concentrations to the Omicron BA.1 subvariant, assessed at Day 14 following initial study vaccination and analyzed by previous vaccine combination received.
Part 2: Neutralizing Antibody (NAb) GMTs to the Omicron BA.5 subvariant expressed as GMTs | Day 28
  Neutralizing antibody (NAb) GMTs to the Omicron BA.5 subvariant, assessed at Day 28 following initial study vaccination.
Part 2: Neutralizing Antibody (NAb) titers to the Omicron BA.5 subvariant expressed as SRRs | Day 28
  SRRs in NAb titer concentrations to the Omicron BA.5 subvariant, assessed at Day 28 following initial study vaccination
Part 2: Neutralizing Antibody (NAb) titers to the ancestral (Wuhan) strain expressed as GMTs | Day 28
  NAb GMTs to the ancestral (Wuhan) strain, assessed at Day 28 following initial study vaccination.

SECONDARY OUTCOMES:
Part 1: MN50 geometric mean titers (GMTs) to the ancestral (Wuhan),and Omicron BA.1 viruses expressed as GMT | Day 0 to Day 240
  MN50 GMTs to the ancestral (Wuhan), and Omicron BA.1 viruses at relevant time points (Days 0, 7, 14, 28, and 240) and analyzed by previous vaccine combination received.
Part 1: MN50 titer concentrations to the ancestral (Wuhan), and Omicron BA.1 viruses expressed as GMFR | Day 7 to Day 240
  MN50 geometric mean fold rise (GMFR) to the ancestral (Wuhan), and Omicron BA.1 viruses at relevant time points (Days 7, 14, 28, and 240) from baseline (Day 0) and analyzed by previous vaccine combination received.
Part 1: MN50 titer concentrations to the ancestral (Wuhan), and Omicron BA.1 viruses expressed as SRRs | Day 7 to Day 240
  SRRs in MN50 titer concentrations to the ancestral (Wuhan), Omicron BA.1, and Omicron BA.5 viruses at relevant time points (Days 7, 14, 28, and 240) and analyzed by previous vaccine combination received.
Part 1: Immunoglobulin G (IgG) antibody levels to the ancestral (Wuhan), Omicron BA.1 and Omicron BA.5 viruses expressed as GMT | Day 0 to Day 240
  Immunoglobulin G (IgG) antibody levels to the ancestral (Wuhan), Omicron BA.1, and Omicron BA.5 viruses at relevant time points (Days 0, 7, 14, 28, and 240) and analyzed by previous vaccine combinations received.
Part 1:IgG antibody levels to the ancestral (Wuhan), Omicron BA.1, and Omicron BA.5 viruses expressed as GMFR | Day 0 to Day 240
  IgG antibody levels to the ancestral (Wuhan), Omicron BA.1, and Omicron BA.5 viruses at relevant time points (Days 0, 7, 14, 28, and 240) and analyzed by previous vaccine combination received.
Part 1: IgG antibody levels to the ancestral (Wuhan), Omicron BA.1 and Omicron BA.5 viruses expressed as SRRs | Day 0 to Day 240
  IgG antibody levels to the ancestral (Wuhan) and Omicron BA.5 viruses at relevant time points (Days 0, 7, 14, 28, and 240) and analyzed by previous vaccine combination received.
Part 1: Human angiotensin-converting enzyme 2 (hACE2) receptor binding inhibition assay to the ancestral (Wuhan), Omicron BA.1, and Omicron BA.5 viruses expressed as GMTs | Day 0 to Day 240
  hACE2 receptor binding inhibition assay to the ancestral (Wuhan), Omicron BA.1, and Omicron BA.5 viruses at relevant time points (Days 0, 7, 14, 28, and 240) and analyzed by previous vaccine combination received.
Part 1: hACE2 receptor binding inhibition assay to the ancestral (Wuhan), Omicron BA.1, and Omicron BA.5 viruses expressed as GMFR | Day 0 to Day 240
  hACE2 receptor binding inhibition assay to the ancestral (Wuhan), Omicron BA.1, and Omicron BA.5 viruses at relevant time points (Days 0, 7, 14, 28, and 240) and analyzed by previous vaccine combination received. Derived/calculated endpoints based on these data will include GMFR.
Part 1: hACE2 receptor binding inhibition assay to the ancestral (Wuhan), Omicron BA.1, and Omicron BA.5 S proteins expressed as SRR | Day 0 to Day 240
  hACE2 receptor binding inhibition assay to the ancestral (Wuhan), Omicron BA.1, and Omicron BA.5 S proteins at relevant time points (Days 0, 7, 14, 28, and 240) and analyzed by previous vaccine combination received. Derived/calculated endpoints based on these data will include SRRs.
Part 1: MN50 GMTs to the to the ancestral (Wuhan) virus expressed as GMT | Day 14
  MN50 GMTs to the ancestral (Wuhan) virus, assessed at Day 14 following initial study vaccination and analyzed by previous vaccine combination received.
Part 1: MN50 GMTs to the to the ancestral (Wuhan) virus expressed as GMFR | Day 14
  MN50 GMFRs to the ancestral (Wuhan) virus at Day 14, from baseline (Day 0) and analyzed by previous vaccine combination received.
Part 1: SRRs in MN50 titer concentrations to the ancestral (Wuhan) virus expressed as SRRs | Day 14
  SRR in MN50 titer concentrations to the ancestral (Wuhan) virus, assessed at Day 14 following initial study vaccination.
Part 1: MN50 GMTs to the Omicron BA.1 subvariant virus expressed as GMT | Day 14
  MN50 GMTs to the Omicron BA.1 subvariant virus, assessed at Day 14 following initial study vaccination and analyzed by previous vaccine combination received.
Part 1: MN50 GMTs to the Omicron BA.1 subvariant virus expressed as GMFR | Day 14
  MN50 GMFRs to the Omicron BA.1 subvariant virus at Day 14, from baseline (Day 0) and analyzed by previous vaccine combination received.
Part 1: MN50 GMTs to the Omicron BA.1 subvariant virus expressed as SRR | Day 14
  SRR in MN50 titer concentrations to the Omicron BA.1 variant virus, assessed at Day 14 following initial study vaccination.
Part 1 and Part 2: Incidence of solicited local and systemic Adverse Events (AEs) | Day 7
  Incidence, duration, and severity of solicited local and systemic AEs for 7 days following vaccination.
Part 1 and Part 2 : Incidence of unsolicited AEs | Day 28
  Incidence, duration, severity, and relationship of unsolicited AEs through 28 days after vaccination.
Part 1 and Part 2 :Incidence and relationship of Medically Attended Adverse Event(s) (MAAEs), Adverse event(s) of Special Interest (AESIs), and Serious Adverse Event(s) (SAEs) | Day 0 to Day 270
  Incidence and relationship of MAAEs, AESIs (predefined list), and SAEs throughout the study
Part 1: IgG Geometric Mean Concentrations (GMCs) to the ancestral (Wuhan), Omicron BA.1, and Omicron BA.5 S proteins expressed as GMFR | Day 0 to Day 240
  IgG GMCs to the ancestral (Wuhan), Omicron BA.1, and Omicron BA.5 S proteins at relevant time points (Days 0, 7, 14, 28, and 240) and analyzed by previous vaccine combination received.
Part 1: IgG GMCs to the ancestral (Wuhan), Omicron BA.1, and Omicron BA.5 S proteins expressed as SRR | Day 0 to Day 240
  IgG GMCs to the ancestral (Wuhan), Omicron BA.1, and Omicron BA.5 S proteins at relevant time points (Days 0, 7, 14, 28, and 240) and analyzed by previous vaccine combination received.
Part 1: GMTs to the ancestral (Wuhan), Omicron BA.1, and Omicron BA.5 S proteins expressed as SRR | Day 0 to Day 240
  GMTs to the ancestral (Wuhan), Omicron BA.1, and Omicron BA.5 S proteins at relevant time points (Days 0, 7, 14, 28, and 240) and analyzed by previous vaccine combination received.
Part 1: GMTs to the ancestral (Wuhan), Omicron BA.1, and Omicron BA.5 S proteins expressed as GMFR | Day 0 to Day 240
  GMTs to the ancestral (Wuhan), Omicron BA.1, and Omicron BA.5 S proteins at relevant time points (Days 0, 7, 14, 28, and 240) and analyzed by previous vaccine combination received.
Part 2: Neutralizing Antibody (NAb) titers to the ancestral (Wuhan) and Omicron BA.5 strains expressed as GMTs | Day 0 to Day 270
  NAb GMTs to the ancestral (Wuhan) and Omicron BA.5 strains at relevant time points (Days 0, 14, 28, 90, 104, 118, and 270) and analyzed by age group (overall, 18 to 54, and ≥ 55 years of age).
Part 2: Neutralizing Antibody (NAb) titers to the ancestral (Wuhan) and Omicron BA.5 strains expressed as GMFRs | Day 0 to Day 270
  NAb GMFR to the ancestral (Wuhan), and Omicron BA.5 strains at relevant time points (Days 14, 28, 104, 118, and 270) from baseline (Day 0 or Day 90) and analyzed by age group (overall, 18 to 54, and ≥ 55 years of age).
Part 2: Neutralizing Antibody (NAb) titers to the ancestral (Wuhan) and Omicron BA.5 strains expressed as SRRs | Day 0 to Day 270
  SRRs in NAb titers to the ancestral (Wuhan) and Omicron BA.5 strains at relevant time points (Days 14, 28, 104, 118, and 270) and analyzed by age group (overall, 18 to 54, and ≥ 55 years of age).
Part 2: IgG GMEUs antibody levels to the ancestral (Wuhan) and Omicron BA.5 S proteins expressed as GMTs | Day 0 to Day 270
  IgG GMEUs to the ancestral (Wuhan) and Omicron BA.5 S proteins at relevant time points (Days 0, 14, 28, 90, 104, 118, and 270) and analyzed by age group (overall, 18 to 54, and ≥ 55 years of age).
Part 2: IgG GMEUs antibody levels to the ancestral (Wuhan) and Omicron BA.5 S proteins expressed as GMFRs | Day 0 to Day 270
  IgG GMEUs to the ancestral (Wuhan) and Omicron BA.5 S proteins at relevant time points (Days 0, 14, 28, 90, 104, 118, and 270) and analyzed by age group (overall, 18 to 54, and ≥ 55 years of age).
Part 2: IgG GMEUs antibody levels to the ancestral (Wuhan) and Omicron BA.5 S proteins expressed as SRRs | Day 0 to Day 270
  IgG GMEUs to the ancestral (Wuhan) and Omicron BA.5 S proteins at relevant time points (Days 0, 14, 28, 90, 104, 118, and 270) and analyzed by age group (overall, 18 to 54, and ≥ 55 years of age).
Part 2:hACE2 receptor binding inhibition assay to the ancestral (Wuhan),and Omicron BA.5 S proteins expressed as GMTs | Day 0 to Day 270
  hACE2 receptor binding inhibition assay GMTs to the ancestral (Wuhan) and Omicron BA.5 S proteins at relevant time points (Days 0, 14, 28, 90, 104, 118, and 270) and analyzed by age group (overall, 18 to 54, and ≥ 55 years of age).
Part 2:hACE2 receptor binding inhibition assay to the ancestral (Wuhan), and Omicron BA.5 S proteins expressed as GMFRs | Day 0 to Day 270
  hACE2 receptor binding inhibition assay GMTs to the ancestral (Wuhan) and Omicron BA.5 S proteins at relevant time points (Days 0, 14, 28, 90, 104, 118, and 270) and analyzed by age group (overall, 18 to 54, and ≥ 55 years of age).
Part 2:hACE2 receptor binding inhibition assay to the ancestral (Wuhan), and Omicron BA.5 S proteins expressed as SRRs | Day 0 to Day 270
  hACE2 receptor binding inhibition assay GMTs to the ancestral (Wuhan) and Omicron BA.5 S proteins at relevant time points (Days 0, 14, 28, 90, 104, 118, and 270) and analyzed by age group (overall, 18 to 54, and ≥ 55 years of age).

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development, Study Director — Novavax, Inc.
Locations (19):
- Australia (19):
  - Paratus Clinical Research Canberra, Bruce, Australian Capital Territory
  - Paratus Clinical Research Western Sydney, Blacktown, New South Wales
  - Emeritus Research, Botany, New South Wales
  - Northern Beaches Clinical Research, Brookvale, New South Wales
  - Paratus Clinical Research Central Coast, Kanwal, New South Wales
  - Australian Clinical Research Network (ACRN), Maroubra, New South Wales
  - AIM Centre (Hunter Diabetes Centre), Merewether, New South Wales
  - Novatrials, Newcastle, New South Wales
  - Holdsworth House Medical Practice, Sydney, New South Whales
  - Paratus Clinical Research Brisbane, Albion, Queensland
  - Core Research Group Pty Ltd, Milton, Queensland
  - Griffith University Clinical Trial Unit, Southport, Queensland
  - Data Health Australia PTY Ltd t/a Austrials, Taringa, Queensland
  - AusTrials Wellers Hill, Wellers Hill, Queensland
  - Clinical Medical and Analytical Excellence (CMAX), Adelaide, South Australia
  - Eastern Health-Box Hill Hospital, Box Hill, Victoria
  - Emeritus Research, Camberwell, Victoria
  - University Hospital Geelong-Barwon Health, Geelong, Victoria
  - Monash Health -Monash Medical Centre, Melbourne, Victoria

REFERENCES:
- [Derived] Bennett C, Rivers EJ, Woo W, Bloch M, Cheung K, Griffin P, Mohan R, Deshmukh S, Arya M, Cumming O, Neville AM, Pardey TM, Plested JS, Cloney-Clark S, Zhu M, Kalkeri R, Patel N, Buchanan A, Marcheschi A, Swan J, Smith G, Cho I, Glenn GM, Walker R, Mallory RM. Immunogenicity and Safety of Heterologous Omicron BA.1 and Bivalent SARS-CoV-2 Recombinant Spike Protein Booster Vaccines: A Phase 3 Randomized Clinical Trial. J Infect Dis. 2024 Jul 25;230(1):e4-e16. doi: 10.1093/infdis/jiad508. PMID 39052718
- [Derived] Bennett C, Woo W, Bloch M, Cheung K, Griffin P, Mohan R, Deshmukh S, Arya M, Cumming O, Neville AM, McCallum Pardey TG, Plested JS, Cloney-Clark S, Zhu M, Kalkeri R, Patel N, Marcheschi A, Swan J, Smith G, Cho I, Glenn GM, Walker R, Mallory RM; Novavax 2019nCoV-311 Study Group. Immunogenicity and safety of a bivalent (omicron BA.5 plus ancestral) SARS-CoV-2 recombinant spike protein vaccine as a heterologous booster dose: interim analysis of a phase 3, non-inferiority, randomised, clinical trial. Lancet Infect Dis. 2024 Jun;24(6):581-593. doi: 10.1016/S1473-3099(24)00077-X. Epub 2024 Mar 6. PMID 38460525